CLINICAL TRIAL: NCT04843436
Title: Post-Market, Non-Randomized, Multicentre PMCF Study to Monitor the Safety and Performance of Symani System in Microsurgical Reconstructive Procedures in a Real Life Setting
Brief Title: PRIMO Post-Market Clinical Follow Up Study
Acronym: PRIMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MMI (Medical Microinstruments, Inc.) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-00031
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Open Surgery; Blood Vessels, Lymphatic Ducts and Nerves; Free Flaps
Keywords: microsurgery; RASM; free flap; lymphatic ducts; Symani

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic Assisted Microsurgery (Experimental): Patients who meet the eligibility criteria for the study and undergo a microsurgical reconstruction using the Symani System according to its indications for use.
  Interventions: Device: Symani Surgical System

INTERVENTIONS:
Device: Symani Surgical System — Robotically Assisted Microsurgery

SUMMARY:
Post Market Clinical Follow up Study aimed to collect clinical data on safety and efficacy of Robotically Assisted System called Symani to perform microsurgery techniques such as anastomosis, suturing and ligation for open surgery procedures on small anatomical structures such as blood vessels, lymphatic ducts and nerves.

DETAILED DESCRIPTION:
PMCF study aimed to monitor the safety, usability, performance and long-term efficacy of Symani. Furthermore, it will permit to detect potential emerging risks related to safety on the basis of clinical evidence through the observation of patients who have undergone microsurgical reconstructions using the Symani Surgical System in the usual setting of standard surgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged >18
* Patients who need a reconstructive procedure and a microsurgical reconstruction is deemed the best option by the plastic, orthopedic or other surgeon in response to a post-oncological, post-traumatic or congenital tissue defect or to treat lymphedema.
* Patients who have been selected by the PI at the Clinical Center as appropriate candidates for treatment with Symani System in accordance with the IFU.
* Subjects who fit the criteria to perform surgery requiring reconstructions using free flaps, replantation, lymphatic reconstructions.
* Subjects who agree to have the surgery and the anaesthesia.
* Subjects who voluntarily decide to participate in this study with the surgery performed with the aid of the Symani System and sign the Informed Consent Form.

Exclusion Criteria:

* Subjects who have bleeding or coagulation disorders in the past or present.
* Any criteria that preclude prolonged anesthesia.
* History of anaphylaxis or severe complicated allergy symptoms.
* Clinically significant cardiovascular, digestive, respiratory, endocrine, or central nervous system disorders or previous mental disorders that may significantly affect the data collection or the ability to comply with the protocol.
* Evidence or history of autoimmune disease or compromised immune system.
* Participation in another clinical trial within 4 weeks prior to participation in the study.
* Subjects belonging to vulnerable populations or ineligible to participate for other reasons by the PI at a Clinical Center.
* Subjects with pacemaker

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 427 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2025-02-06 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Procedure Robotic Success | Procedure
  Ability to complete the surgical task with Symani as intended by the surgeon

SECONDARY OUTCOMES:
Anastomosis time | Procedure
  Time to execute each anastomosis
Intraoperative redo | Procedure
  Intraoperative need to repeat anastomosis
Postoperative redo | 7 days
  Postoperative need to repeat anastomosis
Complications | 30 days
  Major or minor complications
Free Flap/Replantation Failure | 30 days
  Failure of the free flap or replantation
Limb volume reduction (for lymphatic surgery) | 24 weeks
  Limb volume reduction
Warm ischemia time | Procedure
  Time for warm ischemia

CONTACTS AND LOCATIONS:
Overall Officials: Marco Innocenti, Prof., Principal Investigator — Istituto Ortopedico Rizzoli Bologna
Locations (10):
- LKH Salzburg, Universitätsklinik für Mund-, Kiefer- und Gesichtschirurgie, Salzburg, Austria
- Universitair Ziekenhuis Brussel, Brussels, Belgium
- Helsinki University Hospital, Helsinki, Finland
- Germany (3):
  - Klinik für Mund-, Kiefer- und Gesichtschirurgie UKSH Kiel, Kiel
  - BG Kliniken Ludwigshafen, Ludwigshafen
  - Fachklinik Hornheide, Münster
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No